CLINICAL TRIAL: NCT07118748
Title: Dispensing of Antibiotics in Pharmacies for Cystitis According to a Delegation Protocol, Impact of a Decision Support Tool : a Randomised Cluster Trial. PHARIBO: PHarmacy and Resolved Antibiotherapy for Urinary Tract Infections
Brief Title: Dispensing of Antibiotics in Pharmacies for Cystitis According to a Delegation Protocol, Impact of a Decision Support Tool. PHARIBO: PHarmacy and Resolved Antibiotherapy for Urinary Tract Infections
Acronym: PHARIBO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2024/66
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Acute Cystitis
Keywords: cystitis; professional delegation; share decision making; antibiotics
MeSH Terms: conditions — Cystitis

STUDY DESIGN:
Intervention Model Description: open-label, two-arms cluster randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Share making tool decision group (Experimental): woman, between 18 and 65 years, coming to a pharmacy randomized in the experimental group for symptom of acute cystitis without risk of complication
  Interventions: Other: Share making decision tool
- Delegation protocol alone group (Active Comparator): woman, between 18 and 65 years, coming to a pharmacy randomized in the control group for symptom of acute cystitis without risk of complication
  Interventions: Other: Delegation protocol

INTERVENTIONS:
Other: Share making decision tool — the experimental group will apply the delegation protocol, but if the protocol recommends antibiotic therapy, the researchers will propose a shared decision using a specific tool to determine with the patient whether to deliver the antibiotic
  Arms: Share making tool decision group
Other: Delegation protocol — the control group will apply the delegation protocol alone
  Arms: Delegation protocol alone group

SUMMARY:
The purpose of this trial is to demonstrate that when treating acute cystitis without risk of complication, pharmacists may use share Decision Making tool to help patients to better understand the stakes of taking antibiotics and adapt the management of the delegation protocol.

This will select patients in need of antibiotics and preserve the full-capacities of non-treated one.

DETAILED DESCRIPTION:
Each year, in France, more than 2.000.000 patients visit for a acute cystitis. The literature shows that acute cystitis without risk of complication cause pyelonephritis only on really rare situation, but french delegation protocols to pharmacist ask for systematic antibiotic therapy as soon as the diagnostic is made with the only goal to lowering symptomatology. Studies shows that some informed women would like not to take antibiotics while others studies show us that pain-killers could be as effective as antibiotics on case of low symptomatology.

This study will compare a group following only the French protocols for delegating acute cystitis to the pharmacist with a group using the same protocol, but supplementing it with a shared decision-making tool to determine whether, after being informed of the benefits and risks of this treatment, patients still wish to receive an antibiotic. Targeting instead of systematic prescription will reduce antibiotic consumption.

After diagnostic of acute cystitis to a woman between 18 and 65 years, investigators check if they filing all study criteria and ask for authorization to add them to the study. Then they'll act following their group instruction, and get informations (antibiotic prescription or not, patient socio-demographic criteria). Then patients will be followed by telephone on D14 to know if they've take antibiotics and to obtain the following information: AIA scale, O'Connor Scale, Satisfaction scale, if there has been visit to the emergency room or doctor. Antibiotics delivery on pharmacy will be watch by National assurance number of the included patients

ELIGIBILITY:
Inclusion Criteria:

* woman,
* symptom of acute cystitis without risk of complication,
* affiliated to the french public welfare system,
* signed consent.

Exclusion Criteria:

* anomaly of the urinary canal,
* pregnancy, more than 3 cystitis during the last year,
* cancer,
* immunosuppression,
* hemopathy,
* fever,
* back-pain,
* severe renal failure,
* refuse to give consent and previously participate to the study,
* under guardianship.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Dispensing of antibiotic | day 14 after inclusion
  Dispensing of antibiotic for acute cystitis without risk of complication on the 14 days following the first visit to the pharmacy.

SECONDARY OUTCOMES:
Activity Impairment Assessment(AIA) scale | day 14 after inclusion
  5-item ranging from 0 (no impact) to 4 (constant impact). It has no sub-dimensions and allows for an overall assessment (sum of the scores for each item) ranging from 0 (no discomfort/no incapacity) to 20 (total discomfort/ total incapacity).
Satisfaction scale | day 14 after inclusion
  Satisfaction score on a scale from 0 (dissatisfaction) to 10 (total satisfaction)
O'Connor scale | day 14 after inclusion
  16-item scale rated from 1 to 5. Each score is converted to a base of 100 (1=0, 5=100).
  The total average of the items out of 100 determines:
  < 25: Low conflict - the person is probably ready to make a decision. 25-37.5: Moderate conflict - some discomfort may still exist.
  ≥ 37.5: High conflict - the person probably needs help deciding.
Medical consultation | day 14 after inclusion
  Consultations with a doctor or at the emergency room for urinary tract infection and/or possible complications among patients diagnosed with uncomplicated cystitis within two weeks of visiting the pharmacy (telephone survey at two weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No